CLINICAL TRIAL: NCT00503243
Title: A Phase III, Randomized, Multi-Centre, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of SPD476 (Mesalazine) Given Twice Daily (2.4 g/Day) Versus SPD476 Given as a Single Dose (4.8 g/Day) in Subjects With Acute Mild to Moderate Ulcerative Colitis
Brief Title: Safety and Efficacy of SPD476 (Mesalazine) Given Twice Daily (2.4 g/Day) vs SPD476 Given as a Single Dose (4.8 g/Day) in Subjects With Acute Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD476-301; 2004-000733-12 (EudraCT Number)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Drug: Delayed and extended release mesalazine

SUMMARY:
The aim of this study was to investigate the safety and efficacy of SPD476 2.4 g/day given twice daily ([BID] ie 1.2 g/day BID) and SPD476 4.8g/day given QD compared to placebo in subjects with acute, mild to moderate ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed or diagnosis of relapsing (relapsed <= 6 weeks to baseline) mild to moderate ulcerative colitis
* women not of childbearing potential or WOCP who agreed to use an effective contraceptive method

Exclusion Criteria:

* severe ulcerative colitis or relapsed for > 6 weeks prior to baseline
* subjects who had relapsed on maintenance therapy with doses of mesalazine > 2.0 g/day
* subjects with Crohn's disease, proctitis, bleeding disorders or active peptic ulcer disease
* subjects with asthma if they were known to be mesalazine-sensitive
* subjects who were at immediate or significant risk of toxic megacolon
* subjects who had previous resective colonic surgery
* subjects who had moderate or severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2003-09-30 (Actual); Primary Completion 2005-01-17 (Actual); Study Completion 2005-01-17 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in remission (Ulcerative Colitis Disease Activity Index score of <= 1, with scores of 0 for rectal bleeding and stool frequency, and a sigmoidoscopy score reduction of 1 point or more from baseline | 8 weeks

SECONDARY OUTCOMES:
Clinical improvement as defined by a drop of => 3 points from baseline in the overall UC-DAI score | 8 weeks
Change in the UC-DAI score | 8 weeks
Change in symptoms (rectal bleeding and stool frequency) | 2, 4 and 8 weeks
Change in sigmoidoscopic (mucosal) appearance | 8 weeks
Time to withdrawal from the start of study medication | Throughout the study period of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Lichtenstein GR, Kamm MA, Boddu P, Gubergrits N, Lyne A, Butler T, Lees K, Joseph RE, Sandborn WJ. Effect of once- or twice-daily MMX mesalamine (SPD476) for the induction of remission of mild to moderately active ulcerative colitis. Clin Gastroenterol Hepatol. 2007 Jan;5(1):95-102. doi: 10.1016/j.cgh.2006.10.025. PMID 17234558
- See also: FDA-approved label, US only — http://www.lialda.com/Professional/pdf/pi.pdf
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html